CLINICAL TRIAL: NCT05059899
Title: Community WALKing and Home-baSed circuiT tRaining in peOple liviNG With Intermittent Claudication (WALK-STRONG): a Randomised Controlled Feasibility Trial
Brief Title: Home-based Circuit Training for People With Intermittent Claudication
Acronym: WALKSTRONG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coventry University (Other)
Collaborators: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Principal Investigator, Alex Waddell, Principle Investigator, Coventry University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P123339
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication
Keywords: home-based exercise; circuit training; walking
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Home-based circuit and community walking exercise
  Interventions: Behavioral: Exercise group
- Usual care (No Intervention): Usual activity/healthcare

INTERVENTIONS:
Behavioral: Exercise group — The exercise group will receive a 12-week home-based exercise programme, with a wearable activity watch to regulate physical activity behaviour. This group will also receive biweekly telephone calls from the investigator.
  Arms: Exercise group

SUMMARY:
The purpose of the study is to assess the feasibility of undertaking a randomised controlled trial investigating the effectiveness of a 12-week home-based exercise programme for people with intermittent claudication.

DETAILED DESCRIPTION:
30 participants with PAD will be randomised to one of two groups: either exercise or usual care. The 12 week exercise intervention will consist of a home-based circuit programme, including both resistance exercises and walking. This will be combined with promoting free-living walking throughout the rest of the week. Exercise will be regulated via the use of a wearable activity monitor. Biweekly phone calls will address compliance with the intervention. The primary outcomes are feasibility and acceptability, which will be determined after 12 weeks via recruitment and attrition rates, protocol adherence and with participant interviews. Secondary outcomes include changes in pain-free and maximal walking distances with both a graded treadmill test and six-minute walk test, hand grip strength, physical activity behaviour (measured with an accelerometer), quality of life (measured with the SF-36, VascuQol and E5-5D-5L questionnaires) after 12 and 24 weeks. Investigators will also assess changes in markers of inflammation, vascular remodeling, mitochondrial biogenesis and oxidative stress at 12 and 24 weeks. Other outcomes include changes in time spent resting during a six-minute walk test and time to pain cessation following a graded treadmill test at 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ankle/brachial index (ABPI) < 0.9 at rest or a drop of 20mmHg after exercise testing
* Ability to walk independently
* English speaking
* Able to follow instructions
* ≥ 18 years of age

Exclusion Criteria:

* Unable to provide informed consent
* Walking impairment for a reason that is not PAD
* Critical limb ischaemia
* Asymptomatic PAD
* Active cancer treatment
* Severe mental or physical limitations precluding participation safely in the home environment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility assessed via recruitment rate | Will be evaluated after the intervention period (i.e.. 24 weeks after inclusion)
  The investigators will record the number of eligible participants, as well as the number who enroll onto the study.
Intervention feasibility assessed via attrition rate | Will be evaluated after the intervention period (i.e.. 24 weeks after inclusion)
  The investigators will record the number of protocol discontinuations and losses to follow-up.
Intervention feasibility assessed via protocol adherence | Will be evaluated after the intervention period (i.e.. 24 weeks after inclusion)
  The investigators will examine discrepancies between intervention prescription and what is completed.
Intervention acceptability via participant interviews | Will be evaluated after the intervention period (either at 12 week or 24 week follow up)
  One-to-one interviews will be held between an investigator and participant who has either completed the intervention, withdrawn or declined participation, to ask questions regarding the intervention protocol.

SECONDARY OUTCOMES:
12 and 24 week change in six-minute walk distance and pain-free walk distance | Baseline to 12 weeks and 24 weeks
  Change in six-minute and pain-free walk distance after 12 and 24 weeks will be compared to participants randomised to the exercise group vs the usual care group.
12 and 24 week change in pain-free and maximal treadmill walk distance | Baseline to 12 weeks and 24 weeks
  Change in pain-free and maximal treadmill walk distance after 12 and 24 weeks will be compared to participants randomised to the exercise group vs the usual care group.
12 and 24 weeks change in left and right hand grip strength (via hand held dynamometer) | Baseline to 12 weeks and 24 weeks
  Change in left and right hand grip strength after 12 and 24 weeks will be compared to participants randomised to the exercise group vs the usual care group.
12 and 24 week change in physical activity measured by accelerometer data | Baseline to 12 weeks and 24 weeks
  Change in physical activity behaviour at 12 and 24 weeks will be compared to participants randomised to the exercise group vs the usual care group, using accelerometer data.
12 and 24 week change in SF-36 score | Baseline to 12 weeks and 24 weeks
  Change in 36 Item Short Form survey scores at 12 and 24 weeks will be compared to participants randomised to the exercise group vs the usual care group. (Score ranges from 0-100, with higher scores associated with a better outcome).
12 and 24 week change in VascuQol questionnaire score | Baseline to 12 weeks and 24 weeks
  Change in Vascular Quality of Life questionnaire scores at 12 and 24 weeks will be compared to participants randomised to the exercise group vs the usual care group. (Score ranges from 1-7, with higher scores associated with a better outcome).
12 and 24 week change in EQ-5D-5L questionnaire score | Baseline to 12 weeks and 24 weeks
  Change in European Quality of Life Five Dimension questionnaire scores at 12 and 24 weeks will be compared to participants randomised to the exercise group vs the usual care group. (Scores range from 1-5, with lower scores associated with a better outcome).
12 and 24 week change in circulating markers of inflammation | Baseline to 12 weeks and 24 weeks
  Investigators will compare blood sample measures of IL-6, TNF-α, CRP between participants randomised to the exercise group vs the usual care group at 12 and 24 weeks.
12 and 24 week change in circulating markers of vascular remodelling | Baseline to 12 weeks and 24 weeks
  Investigators will compare blood sample measures of VEGF between participants randomised to the exercise group vs the usual care group at 12 and 24 weeks.

OTHER OUTCOMES:
12 and 24 week change in rest times during a six-minute walk test | Baseline to 12 weeks and 24 weeks
  Change in time spent resting during a six-minute walk test after 12 and 24 weeks will be compared to participants randomised to the exercise group vs the usual care group.
12 and 24 week change in pain cessation following a treadmill test | Baseline to 12 weeks and 24 weeks
  Change in time to pain cessation following a treadmill test after 12 and 24 weeks will be compared to participants randomised to the exercise group vs the usual care group.
12 and 24 week changes in walking speed during a six-minute walk test | Baseline to 12 weeks and 24 weeks
  Change in walking speed during a six-minute walk test after 12 and 24 weeks will be compared to participants randomised to the exercise group vs the usual care group.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Waddell, MSc, Principal Investigator — Coventry University
Locations (1):
- Coventry University, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waddell A, Denton F, Powell R, Broom DR, Birkett ST, McGregor G, Harwood AE. "It's put a routine and regimen in my life" - Participant experiences with a programme of community walking and home-based circuit training for intermittent claudication. J Vasc Nurs. 2024 Dec;42(4):276-281. doi: 10.1016/j.jvn.2024.09.003. Epub 2024 Sep 28. PMID 39645388